CLINICAL TRIAL: NCT04989673
Title: Materno-fetal Consequences of Symptomatic Dengue in Pregnant Wowen in French Guiana
Acronym: CMFdeng
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cayenne (Other)
Collaborators: Centre Hospitalier de Kourou (Unknown); Centre Hospitalier de l'Ouest Guyanais (Unknown); Centres de Protection Maternelle Infantile Cayenne, Kourou et Saint-Laurent du Maroni (Unknown); Private physicians Cayenne, Kourou et Saint-Laurent du Maroni (Unknown); Private midwife Cayenne, Kourou et Saint-Laurent du Maroni (Unknown)
Responsible Party: Sponsor
Other Study IDs: CMFdeng
Record Dates: First submitted 2021-07-26; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Dengue; Pregnancy Preterm; Women; Fever; Parturition; Precipitate; Infant, Newborn
Keywords: Symptomatic Dengue; Pregnancy Preterm; Vertical transmission; Fetus; French Guiana
MeSH Terms: conditions — Dengue; Fever | interventions — Surveys and Questionnaires; Data Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tubes of venous blood and or placenta sampling
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Exposed group (GE): Pregnant women with symptomatic dengue fever, confirmed biologically between the presumed date of conception and the date of delivery.
  Interventions: Other: Biological sampling and collection (serum); Other: Biological sampling and collection (placenta); Other: Questionnaire; Other: Data collection
- Unexposed group with fever (GNEF): Pregnant women presenting a febrile syndrome not due to the dengue virus between the presumed date of conception and the date of delivery, excluding malaria, rubella, toxoplasmosis, chickenpox, listeriosis, CMV infection and primary HIV infection.
  Interventions: Other: Biological sampling and collection (serum); Other: Questionnaire; Other: Data collection
- Unexposed group without fever or dengue (GNES): Pregnant women exhibiting neither febrile syndrome nor asymptomatic dengue fever between the presumed date of conception and the date of delivery.
  Interventions: Other: Biological sampling and collection (serum); Other: Questionnaire; Other: Data collection

INTERVENTIONS:
Other: Biological sampling and collection (serum) — Detection of the dengue virus during the next scheduled biological assessment as part of normal pregnancy monitoring (additional tube of blood) among women from GNES and GNEF groups
Other: Biological sampling and collection (placenta) — Detection of dengue virus in the placenta of GE patients (additional tube of placenta)
  Groups: Exposed group (GE)
Other: Questionnaire — Questionnaire on the patient's socio-economic conditions (10-minute interview with the Clinical Research Associate, CRA).
Other: Data collection — Case Report Form will be completed by a Clinical Research Associate (CRA) from the medical file of the patient concerned and of her child at the 3 visits carried out (Pre inclusion V0 or Inclusion V1, Childbirth V2 and Maternity leave V3).

SUMMARY:
Symptomatic dengue virus infection in pregnant women could affect the mother, fetus and the newborn at birth. The risks of postpartum hemorrhage, prematurity and low birth weight are increased in dengue fever. Cases of vertical transmission have been described. This study therefore proposes to quantify these risks in a pregnant woman presenting a clinical picture of dengue fever through a prospective, longitudinal and comparative study.

DETAILED DESCRIPTION:
The main objective of the study is to compare the occurrence of prematurity between women who presented with symptomatic dengue fever and those who did not. However, febrile syndrome is known to be one of the main major risk factors for prematurity whatever its etiology (National College of French Gynecologists and Obstetricians CNGOF, High Authority of Health HAS). Dividing the unexposed group into 2 groups (group without fever or dengue GNES and group with fever not due to the dengue virus GNEF) is a means of observing on the one hand the effects of symptomatic dengue (the combination of effect of fever and the effect of the dengue virus) on the primary endpoint and on the other hand to observe the effects of fever in the context of another infectious pathology on the primary endpoint. This split also makes it easy to control the number of patient enrollments in each unexposed group.

This study protocol is only interested in investigating the impact of symptomatic dengue fever in pregnant women.

Primary objective: Compare the prematurity rate of the woman with symptomatic dengue fever (exposed group: GE) during her pregnancy compared to the woman who had neither fever nor infection with the dengue virus during her pregnancy (unexposed group without fever: GNES).

Secondary objectives:

* Describe the clinical pictures of symptomatic dengue fever in pregnant women;
* Compare the proportion of rates of prematurity, threat of premature delivery, spontaneous miscarriage, pre-eclampsia, eclampsia and delivery haemorrhage between the GE / GNES group and between the GE / GNEF group ( pregnant women who presented with dengue GE, those who had neither fever nor dengue during their pregnancy GNES and those who presented a fever not due to the dengue virus GNEF);
* Compare the proportion of MFIU and hypotrophy of newborns born to mothers between the GE / GNES group and between the GE / GNEF group;
* Describe the clinical and biological pictures of newborns at birth of mothers who presented with symptomatic dengue fever during their pregnancy (GE)
* Describe the morphological, biometric and velocimetric abnormalities of obstetric doppler ultrasounds of pregnant women who presented with dengue fever during their pregnancy (GE).
* Check for the presence of the dengue virus in the placenta of pregnant women who have had dengue fever during their pregnancy (GE).
* Constitute a direct biological collection (serums, placentas) used for the research of the dengue virus.

Epidemiological, etiological exposed-unexposed, multicentric, dynamic and contemporary with biological collection

ELIGIBILITY:
* Exposed group (GE)

Inclusion Criteria:

* presenting a symptomatic dengue fever, confirmed biologically between the presumed date of conception (date determined after the first trimester dating ultrasound) and the date of delivery.

Non inclusion Criteria:

* not presenting biologically confirmed dengue fever;
* with asymptomatic dengue fever between the presumed date of conception and the date of delivery.

  * Unexposed group with fever (GNEF)

Inclusion Criteria:

* presenting an infectious syndrome not due to the dengue virus between the presumed date of conception (date determined after the ultrasound dating of the first trimester) and the date of delivery.

Non inclusion Criteria:

* presenting with an infectious syndrome in the context of rubella (before 18 weeks), chickenpox, malaria, listeriosis, toxoplasmosis, primary HIV infection and CMV infection.

Exclusion Criteria:

* Person included in the study with biologically confirmed dengue fever (symptomatic or not) between the date of inclusion and the date of delivery.

  * Unexposed group without fever or dengue (GNES)

Inclusion Criteria:

* Having neither fever (above 38.5 ° C for more than 48 hours) nor dengue confirmed biologically (symptomatic or not) since the beginning of pregnancy.

Non inclusion criteria:

* Having presented a febrile syndrome (fever above 38.5 ° C for more than 48 hours) or dengue fever confirmed biologically (symptomatic or not) since the beginning of pregnancy.

Exclusion criteria:

People included in the study,

* with biologically confirmed dengue fever (symptomatic or not) between the date of inclusion and the date of delivery;
* having presented a febrile syndrome (fever above 38.5 ° C for more than 48 hours) between inclusion and childbirth.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 628 (Actual)
Dates: Start 2012-07-11 (Actual); Primary Completion 2015-02-12 (Actual); Study Completion 2015-07-11 (Actual)

PRIMARY OUTCOMES:
Prematurity rate | 9 months maximum
  The prematurity rate of each group will be assessed according to the WHO definition: a preterm birth is a birth occurring before the 37th week of amenorrhea and after the 22nd week of amenorrhea of a living fetus of at least equal weight at 500 g. This judgment criterion will be measured by the physician or midwife in charge of the patient, and reported on the RIG and the delivery book of the service. The date of delivery will be determined based on the 1st trimester dating ultrasound. The newborn will be examined by the midwife or pediatrician on the ward and weighed within half an hour after birth. A distinction will be made between medically induced premature delivery (reasons given) and spontaneous.

SECONDARY OUTCOMES:
Threatened Premature Delivery (PAD) rate in each group | 9 months maximum
  The threat of premature delivery is a pathology associating cervical changes and regular and painful uterine contractions occurring between 22 and 36 weeks of amenorrhea + 6 days (HAS).
  Cervical changes will be assessed by endovaginal ultrasound of the cervix on at least 1 of the following criteria:
  * neck length less than or equal to 25mm
  * funnel opening or expansion of the internal orifice of the neck
  * protrusion of amniotic membranes in the cervix.
  The close and regular frequency of uterine contractions (generalized and intermittent hardening of the uterus lasting 30 to 60 seconds) will be objectified by a tocographic recording: at least 3 contractions in 30 minutes. The pain will be assessed by the patient with the possible help of the visual analogue scale (VAS> = 5).
Fetal hypotrophy rate | 9 months maximum
  Fetal hypotrophy corresponds to a biometry below the 10th percentile according to the growth curve of the French College of Fetal Ultrasound (CFEF).
  The diagnosis is based on the measurement during an obstetric ultrasound of the biparietal diameter, head circumference (PC), abdominal diameter, abdominal perimeter (PA) and femoral length (FL).
  The fetal weight is estimated according to the Hadlock formula [46] log10 EPF = 1.326 + 0.0107 PC + 0.0438 PA + 0.158 LF - 0.00326 (PA x LF).
Low birth weight | 9 months maximum
  The low birth weight corresponds to a birth weight below the 10th percentile for the term on the CFEF curve.
  The weight will be measured within half an hour after giving birth.
Postpartum hemorrhage rate | 9 months maximum
  corresponds to a loss of blood of more than 500 ml within 24 hours between birth and leaving the maternity hospital.
  This criterion will be measured by midwives or nurses in the operating room (double collection bag: one for amniotic fluid and the other for blood loss). In postpartum, the loss is estimated daily by the midwives or the physician.
Rate of preeclampsia | 9 months maximum
  Pre-eclampsia is de novo hypertension (SBP> = 140 mmHg or ADP> 90 mmHg) in the second part of pregnancy, with the onset of proteinuria greater than 300 mg / 24h or onset of proteinuria in a woman with chronic hypertension. The hypertension will be objectified on at least two blood pressure measurements in a patient lying down and calm for at least 5 minutes or on a blood pressure holter over 24 hours with a cuff adapted to the body of the patient. Chronic hypertension corresponds to a patient on antihypertensive medication. Proteinuria is defined as the pathological elimination in the urine of a quantity of protein greater than 80 mg / day. The 24-hour urine collection for proteinuria can be done in a hospital setting or on an outpatient basis.
Rate of eclampsia | 9 months maximum
  Eclampsia is defined as the occurrence of seizures, either in the 2nd part of pregnancy, or during childbirth, or in the first 48 hours postpartum, in a woman with preeclampsia.
  The occurrence of convulsions in the patient must be validated by a physician or a midwife.
Rate of fetal death in utero | 9 months maximum
  Fetal death from 22 weeks of amenorrhea. Death will be confirmed by the absence of cardiac activity on obstetric Doppler ultrasound.
Spontaneous abortion rate | 9 months maximum
  Early: before 16 SA Late: between 16 and 22 SA. The death of the fetus will be confirmed by examination by the physician or midwife. It should be verified that this is not a voluntary abortion or that he has had medication or a triggering event.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel CARLES, Principal Investigator — Centre Hospitalier de Saint-Laurent du Maroni
Locations (1):
- General Hospital of Cayenne, Cayenne, French Guiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Basurko C, Carles G, Youssef M, Guindi WE. Maternal and fetal consequences of dengue fever during pregnancy. Eur J Obstet Gynecol Reprod Biol. 2009 Nov;147(1):29-32. doi: 10.1016/j.ejogrb.2009.06.028. Epub 2009 Jul 24. PMID 19632027
- [Background] Carles G, Peiffer H, Talarmin A. Effects of dengue fever during pregnancy in French Guiana. Clin Infect Dis. 1999 Mar;28(3):637-40. doi: 10.1086/515144. PMID 10194092
- [Background] Carles G, Talarmin A, Peneau C, Bertsch M. [Dengue fever and pregnancy. A study of 38 cases in french Guiana]. J Gynecol Obstet Biol Reprod (Paris). 2000 Dec;29(8):758-762. French. PMID 11139712
- [Result] Basurko C, Everhard S, Matheus S, Restrepo M, Hilderal H, Lambert V, Boukhari R, Duvernois JP, Favre A, Valmy L, Nacher M, Carles G. A prospective matched study on symptomatic dengue in pregnancy. PLoS One. 2018 Oct 3;13(10):e0202005. doi: 10.1371/journal.pone.0202005. eCollection 2018. PMID 30281605
- [Result] Basurko C, Matheus S, Hilderal H, Everhard S, Restrepo M, Cuadro-Alvarez E, Lambert V, Boukhari R, Duvernois JP, Favre A, Nacher M, Carles G. Estimating the Risk of Vertical Transmission of Dengue: A Prospective Study. Am J Trop Med Hyg. 2018 Jun;98(6):1826-1832. doi: 10.4269/ajtmh.16-0794. Epub 2018 Apr 19. PMID 29692297